CLINICAL TRIAL: NCT03128697
Title: Clinical Evaluation to Improve Obesity Intervention Prescription: Functional Foods as a Potential Solution for Individuals With a Low Satiety Quotient Phenotype?
Brief Title: Impact of a Satiating Diet in Obese Men With a Low Satiety Phenotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Angelo Tremblay, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MOP-68858
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Appetite Disorders
Keywords: Obesity; Satiety quotient; Appetite control; Weight loss; Satiety phenotype; Functional food
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Satiating diet-Low satiety phenotype (Experimental): Low satiety phenotype subjects who were submitted to the experimental diet (satiating diet) for a 16-week period.
  Interventions: Behavioral: Satiating diet
- Satiating diet-High satiety phenotype (Experimental): High satiety phenotype subjects who were submitted to the experimental diet (satiating diet) for a 16-week period.
  Interventions: Behavioral: Satiating diet
- Control diet-Low satiety phenotype (Active Comparator): Low satiety phenotype subjects who were submitted to the control diet (based on the Canadian Food Guide) for a 16-week period.
  Interventions: Behavioral: Control diet
- Control diet-High satiety phenotype (Active Comparator): High satiety phenotype subjects who were submitted to the control diet (based on the Canadian Food Guide) for a 16-week period.
  Interventions: Behavioral: Control diet

INTERVENTIONS:
Behavioral: Satiating diet
  Arms: Satiating diet-High satiety phenotype; Satiating diet-Low satiety phenotype
Behavioral: Control diet
  Arms: Control diet-High satiety phenotype; Control diet-Low satiety phenotype

SUMMARY:
The global research project was organized as a clinical process starting with an evaluation aiming at the determination of a diagnosis pertaining to the degree of satiety signal capacity. It was extended by a phase of metabolic and behavioural characterization to better understand the clinical condition of the patients. The main part of the program was a weight loss intervention that was focused on high satiating foods. Finally, the process was completed by an evaluation allowing to determine the impact of the intervention on the metabolic and behavioural conditions of the patients.

DETAILED DESCRIPTION:
Dietary restriction, being prescribed as low and very low calorie diets, has been largely used as a strategy of dietary management of obesity. Beyond the fact that these diets fully respect the first law of thermodynamics, they are also rather easy to supervise and they offer a guarantee of substantial weight loss to compliant patients. Dietary restriction strategies also carry important limitations which include their failure to take into account appetite sensations of the obese patient. This point is important since it dictates the extent to which the patient can tolerate his/her dietary regimen without hunger over time as well as its related body weight loss. In this regard, experimental and clinical data show that weight regain up to initial body weight and even more occurs over years after a diet-induced weight loss. Moreover, evidence also revealed that restraint behaviour is difficult to maintain over time and that a decrease in this behaviour is related to weight gain on a long term basis. The challenge thus becomes the search of a strategy that can promote a substantial spontaneous energy deficit without significantly altering hunger and satiety levels as well as their related well-being. Up to now, the only approach which emerges as having the potential to respect these two criteria is the design of functional foods, i.e. foods with sufficient satiety-promoting properties to compensate for the enhancing effect of body fat loss on appetite. The food specialists can rely on a catalogue of functional ingredients that can be used to prepare functional menus in order to improve the regulation of energy balance and body weight stability in individuals prone to obesity. As described above, this issue would be particularly relevant for obese individuals displaying a low satiety phenotype, i.e. individuals experiencing difficulty to match energy intake to expenditure in a context promoting excess food intake.

The objectives of this study were to characterize obese men displaying the low satiety phenotype (metabolic and behavioral characteristics) and to determine the impact of highly satiating foods on body weight loss, satiety feelings and compliance in this population.

EXPERIMENTAL DESIGN

Recruitment of subjects and satiety phenotype determination

Each patient referred by a physician was contacted by phone and a first screening interview was performed to validate the inclusion criteria. After recruitment, every subject was met to read and sign the letter of consent as well as to discuss every aspect of the program about which he might have some questions. We took advantage of this brief meeting to measure height, body weight and waist circumference to determine BMI and to estimate the level of abdominal fat.

This phase also included a 2-hour session of evaluation in order to determine satiety signal capacity (SQ). At the end of this session, each subject completed the Three-Factor Eating Questionnaire with the specific preoccupation to measure cognitive dietary restraint as an exclusion criterion. The information collected in this first phase of testing was used to subsequently classify subjects on the basis of their satiety signal capacity (low SQ vs normal/high SQ). Subjects not selected to participate in the next phase of the project received, in addition to their health report, a free dietary consultation focusing on the adoption of healthy behaviours. This first phase of testing allowed to rank order subjects on the basis of their score obtained with the satiety quotient. Seventy participants were selected to participate in the study

Initial metabolic and behavioural characterization (Time 0)

This phase of testing began by a standard medical examination performed by the physician of our research team several days before the main testing session. This permitted to identify potential illnesses influencing appetite control and to evaluate the general health condition of each subject. In order to evaluate the reproducibility over time of the satiety quotient determination and to ascertain the status of subjects determined at the initial evaluation, the standardized breakfast test meal was repeated. However, this test was performed in a session of longer duration that allowed to characterize metabolic and behavioural factors associated with a low/high satiety capacity. The measurements included in this phase of testing were used as baseline measurements for the next phase of this project.

Intervention study

The 70 participants were randomly assigned to either a weight loss program consisting of a highly satiating diet (n=35) (low to moderate in fat (30-35%), high in fibres (> 25g/day), high protein (20-25% of total energy intake) and including 45-50% energy as carbohydrate mainly provided by foods with low glycemic index and adequate to slightly increased vitamin and mineral intakes) which is expected to induce a spontaneous energy deficit or a diet supervision based on the guidelines concordant with the Canadian Food Guide (n=35) (10-15, 55-60 and 30% energy as protein, carbohydrate, and lipid, respectively). For statistical analysis, 4 subgroups have been created based on the SQ classification: 1) low SQ, high satiating diet 2) low SQ, conventional healthy diet, 3) normal/high SQ, high satiating diet, 4) normal/high SQ, conventional healthy diet. This experimental environment thus corresponded to a two by two factorial design in which the two independent variables are SQ and diet. Participants were encouraged to comply with the diets for a 16-week period even if a resistance to weight loss (i.e weight maintenance during one month) was observed during the protocol.

Final metabolic and behavioural characterization (Post-tests; week 16)

All the measurements performed at Time 0 were repeated immediately after the 16-week intervention period for each of the four subgroups of subjects.

POTENTIAL OUTCOME AND FUTURE PERSPECTIVES

The main conceptual outcomes of this were: 1) the characterization of factors implicated in different satiety signal capacities; 2) the investigation of the role of individual capacity of satiety signal in body weight loss and diet compliance, and 3) the determination of the impact of functional menus promoting satiety to compensate for the low spontaneous satiety level in some obese individuals. In addition, this project provided clinical and economical outcomes. Indeed, it represented the first study documenting the weight-reducing impact of a healthy diet based on foods whose functionality have been upgraded by food design. If this project confirms that such a diet can promote weight loss without restriction, but while rather being associated with well-being, this will be a major gain for clinical nutritionists who have up to now unsuccessfully try to counteract the obesity epidemic and who have to deal with consumers who primarily request palatable foods instead of a priori focusing on healthy food. From an economical standpoint, this program will be a reference source of validation for the industry seeking justifications and claims to promote healthy foods facilitating body weight control.

ELIGIBILITY:
Inclusion Criteria:

* aged between 30 and 50 years
* obese (BMI between 30 and 40 kg/m2)
* overall good health

Exclusion Criteria:

* Participants taking medication which could influence appetite sensations (hormones, tranquillizers such as chlorpromazine and benzodiazepin, lithium carbonate for bipolar disorders, cyproheptadine, antihistaminic, serotonin antagonist, sulfonylurea and glucocorticoids)
* Type 2 diabetic patients treated with insulin
* Large body weight fluctuations (>4 kg over the last two months)
* High level of restraint behaviour (score > 10 as measured with the Three Factor Eating Questionnaire)
* Performing more than 3 x 30 minutes/week of physical activity.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2008-09-30 (Actual); Study Completion 2008-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline body weight at 16 weeks | Pre (Week 0)- and post-intervention (after 16 weeks)
  Body weight (kg)
Change from baseline satiety responsiveness (satiety quotients) at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Measured by a standardized breakfast test meal using visual analogue scales for 4 appetite sensations (hunger, desire to eat, fullness and prospective food consumption) (mm/100kcal)

SECONDARY OUTCOMES:
Change from baseline BMI at 16 weeks | Pre- and post-intervention (week 0 and 16)
  kg/m2
Change from baseline waist circumference at 16 weeks | Pre- and post-intervention (week 0 and 16)
  cm
Change from baseline resting blood pressure at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmHg
Change from baseline resting heart rate at 16 weeks | Pre- and post-intervention (week 0 and 16)
  beat/min
Change from baseline resting energy expenditure at 16 weeks | Pre- and post-intervention (week 0 and 16)
  kcal/day
Change from baseline fat mass at 16 weeks | Pre- and post-intervention (week 0 and 16)
  kg
Change from baseline lean body mass at 16 weeks | Pre- and post-intervention (week 0 and 16)
  kg
Change from baseline percent fat mass at 16 weeks | Pre- and post-intervention (week 0 and 16)
  percent (%)
Change from baseline spontaneous energy intake at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Measured following an ad-libitum buffet-type meal (kcal)
Change from baseline daily energy intake at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three-day dietary record (kcal/day)
Change from baseline diet quality (macronutrient composition) at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three-day dietary record (% carbohydrates, proteins and lipids)
Change from baseline appetite sensations at 16 weeks (desire to eat, fullness, hunger and prospective food consumption) | Pre- and post-intervention (week 0 and 16)
  Measured following an ad-libitum buffet-type meal (0-150 mm).
Change from baseline binge eating tendencies at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Binge Eating Scale (possible score between 0-46)
Change from baseline distress-related body esteem at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Body Esteem Scale (possible score between 0-92)
Change from baseline cognitive restraint at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three Factor Eating Questionnaire (possible score between 0-21)
Change from baseline flexible restraint at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three Factor Eating Questionnaire (possible score between 0-7)
Change from baseline rigid restraint at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three Factor Eating Questionnaire (possible score between 0-7)
Change from baseline disinhibition at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three Factor Eating Questionnaire (possible score between 0-16)
Change from baseline susceptibility for hunger at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Three Factor Eating Questionnaire (possible score between 0-14)
Change from baseline depression symptoms at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Beck Depression Inventory (possible score between 0-63)
Change from baseline anxiety symptoms at 16 weeks | Pre- and post-intervention (week 0 and 16)
  State-Trait Anxiety Inventory (possible score between 20-80)
Change from baseline level of stress at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Perceived Stress Scale (possible score between 0-40)
Change from baseline sleeping quality at 16 weeks | Pre- and post-intervention (week 0 and 16)
  Pittsburgh Sleep Quality (possible score between 0-21)
Change from baseline fasting blood glucose at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood insulin at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood leptin at 16 weeks | Pre- and post-intervention (week 0 and 16)
  ng/ml
Change from baseline fasting blood cortisol at 16 weeks | Pre- and post-intervention (week 0 and 16)
  nmol/L
Change from baseline fasting blood total cholesterol at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood HDL-cholesterol at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood LDL-cholesterol at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood phospholipids at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood triglycerides at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood LDL-apolipoprotein at 16 weeks | Pre- and post-intervention (week 0 and 16)
  mmol/L
Change from baseline fasting blood free T4 at 16 weeks | Pre- and post-intervention (week 0 and 16)
  nmol/L
Change from baseline fasting blood total T3 at 16 weeks | Pre- and post-intervention (week 0 and 16)
  nmol/L
Change from baseline awakening cortisol response at 16 weeks (T0) | Pre- and post-intervention (week 0 and 16)
  Determined from salivary samples taken at the time of awakening (ug/dl)
Change from baseline awakening cortisol response at 16 weeks (T15min) | Pre- and post-intervention (week 0 and 16)
  Determined from salivary samples taken 15 minutes after the awakening (ug/dl)
Change from baseline awakening cortisol response at 16 weeks (T30min) | Pre- and post-intervention (week 0 and 16)
  Determined from salivary samples taken 30 minutes after the awakening (ug/dl)
Change from baseline awakening cortisol response at 16 weeks (T60min) | Pre- and post-intervention (week 0 and 16)
  Determined from salivary samples taken 60 minutes after the awakening (ug/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Tremblay, PhD, Principal Investigator — Laval University; Drapeau Vicky, PhD, Study Director — Laval University
Locations (2):
- Canada (2):
  - Laval University, Québec
  - Laval Hospital, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drapeau V, Blundell J, Gallant AR, Arguin H, Despres JP, Lamarche B, Tremblay A. Behavioural and metabolic characterisation of the low satiety phenotype. Appetite. 2013 Nov;70:67-72. doi: 10.1016/j.appet.2013.05.022. Epub 2013 Jun 20. PMID 23792908
- [Result] Filiatrault ML, Chaput JP, Drapeau V, Tremblay A. Eating behavior traits and sleep as determinants of weight loss in overweight and obese adults. Nutr Diabetes. 2014 Oct 20;4(10):e140. doi: 10.1038/nutd.2014.37. PMID 25329602
- [Result] McNeil J, Drapeau V, Gallant AR, Tremblay A, Doucet E, Chaput JP. Short sleep duration is associated with a lower mean satiety quotient in overweight and obese men. Eur J Clin Nutr. 2013 Dec;67(12):1328-30. doi: 10.1038/ejcn.2013.204. Epub 2013 Oct 16. PMID 24129360